CLINICAL TRIAL: NCT01803997
Title: Pink and Dude Chef Afterschool Cooking Program: Improving Food Knowledge and Skills in Middle School Students
Brief Title: Pink and Dude Chef
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GFHNRC216
Record Dates: First submitted 2012-12-21; First posted 2013-03-04 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Child Nutrition; Fruit and Vegetable Intake; Healthy Food Choice; Healthy Food Preparation
Keywords: Child; Nutrition; resonance Raman spectroscopy; Fruit & Vegetable; Children Cooking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STRIDE (Other): 12 cooking classes offered over 6 weeks (approximately 2 classes/week)
  Interventions: Behavioral: Pink and Dude Chef Afterschool Cooking Program
- SPARK (Other): 12 physical activity classes offered over 6 weeks (approximately 2 classes/week)
  Interventions: Behavioral: Pink and Dude Chef Afterschool Cooking Program

INTERVENTIONS:
Behavioral: Pink and Dude Chef Afterschool Cooking Program — 12 educational cooking classes: two classes per week for six weeks (2 hours each)

SUMMARY:
The purpose of the study is to evaluate an afterschool program to teach nutrition through basic cooking skills. This after school extracurricular program increases the students' confidence, knowledge, and skills for cooking as one of the first steps for dietary improvement. In addition to the life lessons students learn during this class, they gain self-confidence and become self-sufficient culinary experts that are capable of educating their siblings, parents, and social circles. This research project will test the impact this program has on nutritional knowledge, culinary efficacy, and nutritional choices made in and out of the home. The Pink and Dude Chef Afterschool Cooking Program was developed through STRIDE (Science through Translational Research in Diet and Exercise at California Polytechnic state University (Cal Poly) in San Luis Obispo, CA.

Hypothesis: Middle school students participating in the Pink and Dude Chef afterschool cooking program will increase nutritional knowledge, culinary efficacy, motivation to eat fruits and vegetables, and fruit and vegetable intake compared to an attention control group.

ELIGIBILITY:
Inclusion Criteria:

* Middle school aged child with parent willing to partcipate
* Ability to partipate in an afterschool program

Exclusion Criteria:

* Less or greater than middle school aged

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Questionnaire on nutritional knowledge, culinary efficacy, and motivation to eat fruit and vegetables | 6 weeks
  Baseline and post intervention measurements through questionnaires.
Palm scans (resonance Raman spectroscopy) to measure cartenoids (indicator of vegetable and fruit intake). | 6 weeks
  Baseline and post intervention scans.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Grand Forks Human Research Nutrition Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Derived] Casperson SL, Sieling J, Moon J, Johnson L, Roemmich JN, Whigham L. A mobile phone food record app to digitally capture dietary intake for adolescents in a free-living environment: usability study. JMIR Mhealth Uhealth. 2015 Mar 13;3(1):e30. doi: 10.2196/mhealth.3324. PMID 25775506